CLINICAL TRIAL: NCT02379507
Title: DEC033 Study Product for Mild to Moderate Eczema An Open-label, Adaptive-design Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicus Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DECI1200
Record Dates: First submitted 2015-01-13; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-01

CONDITIONS: Eczema
Keywords: mild to moderate
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DEC033 Study Product (Experimental): Apply twice a day
  Interventions: Other: DEC033 Study Product

INTERVENTIONS:
Other: DEC033 Study Product — Apply twice daily

SUMMARY:
This open-label, adaptive design study was designed to determine the efficacy of the study product in the treatment of eczema which would be assessed by the reduction of the appearance of skin lesions and symptoms associated such as itching, scaling and redness.

DETAILED DESCRIPTION:
Eczema is an inflammatory skin disease characterized by itchy red rashes commonly found in the elbows or behind the knees. Eczema lesions may appear as collection of fluid in the skin (vesicles) or as gross thickening of the skin (lichenification) with redness. It is also associated with crusting, scaling, cracking, and swelling of the skin. Usually, it does not need medical treatment. However, a more severe form of eczema is referred to as atopic eczema or atopic dermatitis which occurs in childhood or early adulthood. The overall prevalence of this condition in Northern Europe is 15-20% of children aged 7-18 years. Atopic eczema greatly affects the quality of life of the individuals and in fact accounts for the highest scores when compared with other dermatological diseases. A child with eczema experiences itch and sleep disturbances, ostracism by other children, the need for special clothing and bedding, avoidance of physical activities such as swimming and the need for frequent application of ointments.

Eczema is commonly treated with antihistamine pills and creams or ointments. Antihistamines and steroid creams control the itching and rash caused by severe eczema. It is also recommended that the skin be well lubricated to prevent it from becoming dry. A systematic review of randomized clinical trials on atopic eczema summarized the interventions for treating the condition which include pharmacological drug type (topical steroids), similar intervention type (dietary measures) or convenience (non-pharmacological treatments).

Shea butter, which contains stearic acid, linoleic acid, and catechins (antioxidants), is processed from nut of the Vitellaria paradoxa tree. It is traditionally used as lotion for the skin and hair as it is considered an emollient and skin conditioning agent. It has also been of importance in soothing arthritic pains, reducing swelling, treating skin problems, and as antiseptic for wounds. Shea butter is also found in topical formulations used for inflammatory dermatoses such as psoriasis and atopic dermatitis. Shea butter consists of triterpene cinnamates and acetates and these were found to have anti-inflammatory activity which can help in the reduction of edema associated with eczema. Human clinical studies have demonstrated shea butter as skin aging treatment which regenerates skin and gives smoother, clearer skin. Wrinkles from photoaging were also diminished. Another trial showed that shea butter has cicatrizing action in 70% of cases of hand dermatitis, sun burns and scars. A cream with shea butter was also demonstrated to promote good moisturization of the skin compared to placebo.

Macadamia nut oil is one of the most heart-friendly oils. It contains vitamin E, omega-3, omega-6, oleic, linoleic, and palmitoleic acids. Macadamia oil decreases low density lipoprotein levels and increases high density lipoprotein levels thus reducing risk of heart diseases. There are various benefits of macadamia oil on skin. It provides moisturization and anti-aging effects. Palmitoleic acid, which is commonly found in the skin, decreases as people age. Macadamia oil helps replace the lost compound to maintain youthful skin. Blemishes and scars are also removed with the help of macadamia oil. It has anti-inflammatory activity and antioxidant effects thus reducing free radicals on the skin and providing healing of skin conditions such as sunburns.

This open-label, adaptive design study was designed to determine the efficacy of the study product in the treatment of eczema which would be assessed by the reduction of the appearance of skin lesions and symptoms associated such as itching, scaling and redness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female ≥ 18 and ≤ 70 years of age.
* Body mass index (BMI) ≥ 20 and ≤ 35 kg/m2.
* Subjects with mild to moderate eczema; determined at screening visit.
* Judged by the Investigator to be in general good health on the basis of medical history.
* Agree to use the Study-supplied cleanser and moisturizer as the only body cosmetic applied to irritated skin.
* Agree to stop all medications and supplements during the entire length of the study
* Females of child bearing potential must agree to use appropriate birth control methods during the entire study period.
* Agree not to initiate any new exercise or diet programs during the entire study period.
* Agree not to change their current diet or exercise program during the entire study period.
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.

Exclusion Criteria:

* Clinically significant renal, hepatic, endocrine (including diabetes mellitus), cardiac, pulmonary, pancreatic, neurologic, hematologic, or biliary disorder.
* Known allergy or sensitivity to Herbal products.
* History or presence of cancer in the prior two years, including any skin cancer or suspicious lesions.
* Recent history of alcoholism (within 12 months) or strong potential for alcohol or substance abuse.
* Participation in a clinical study with exposure to any non-registered drug product within 30 days prior.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk. Including subjects who are Bed or wheelchair-bound.
* Pregnant, lactating, or unwilling to use adequate contraception during the duration of the study.
* Smoking - must be nonsmoker for at least 12 weeks prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Symptoms of Itching, Scaling, and Redness measured by Visual Analog Scale (VAS) | 30 days
  Subjects completed the Visual Analog Scale for eczema symptoms - itching, scaling, and redness.

SECONDARY OUTCOMES:
Size and Severity of Eczema Lesions measured by Dermatologic Assessments | 30 days
  Dermatologic assessments for severity and size of lesions and Severity Scoring of Atopic Dermatitis (SCORAD) were assessed by a practitioner in the clinic.